CLINICAL TRIAL: NCT04547907
Title: Comparing the Efficacy of Nab-PHP and TCbHP in Neoadjuvant Therapy for HER2-positive Early Breast Cancer, A Multicenter, Randomized, Phase III Clinical Trial
Brief Title: A Comparison of Nab-PHP and TCbHP Efficacy in Neoadjuvant Therapy for HER2-positive Early Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-006
Record Dates: First submitted 2020-08-29; First posted 2020-09-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer,HER2-positive

STUDY DESIGN:
Intervention Model Description: An open-label, multicenter, randomized controlled phase III clinical study. Neoadjuvant chemotherapy with 6*nab-PHP regimen (experimental group): 344 subjects.
  Neoadjuvant chemotherapy with 6*TCbHP regimen (control group): 344 subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-PHP (Experimental): Nab-paclitaxel + trastuzumab+ patuzumab
  Interventions: Drug: Nab-paclitaxel+ trastuzumab+ patuzumab
- TCbHP (Active Comparator): Docetaxel + carboplatin + trastuzumab + patuzumab
  Interventions: Drug: Docetaxel+ carboplatin+ trastuzumab + patuzumab

INTERVENTIONS:
Drug: Nab-paclitaxel+ trastuzumab+ patuzumab — Nab-paclitaxel 125mg/m2 (days 1, 8, 15) + Trastuzumab (initial loading dose of 8 mg/kg, subsequent maintenance dose of 6 mg/kg) + Pertuzumab (initial loading dose of 840mg, subsequent maintenance dose of 420mg), every 21 days constitute a cycle.
  Other Names: nab-PHP regimen group
  Arms: nab-PHP
Drug: Docetaxel+ carboplatin+ trastuzumab + patuzumab — Docetaxel 75 mg/m2(day 1) + Carboplatin (AUC=6) (day 1) + Trastuzumab (initial loading dose of 8 mg/kg, subsequent maintenance dose of 6 mg/kg) + Pertuzumab (initial loading dose of 840mg, subsequent maintenance dose of 420mg), every 21 days constitute a cycle.
  Other Names: TCbHP regimen group
  Arms: TCbHP

SUMMARY:
The aim of this study is to evaluates the efficacy of weekly nab-paclitaxel monotherapy compared to the standard regimen of docetaxel plus carboplatin, both supplemented with trastuzumab and pertuzumab, as neoadjuvant therapies for HER2-positive breast cancer.

DETAILED DESCRIPTION:
In order to compare the effects of nab-PHP and TCbHP chemotherapy regimens in the neoadjuvant treatment of HER2-positive breast cancer, this study randomly divided patients who met the inclusion criteria into 2 groups through a randomized control regimen： the neoadjuvant chemotherapy with 6*nab-PHP regimen group (experimental group): nab-paclitaxel 125mg/m2 on days 1, 8, and 15 every 21 days as one cycle; 6*TCbHP regimen (control group): docetaxel 75 mg/m2 + carboplatin (AUC=6) on day 1. Both groups will receive trastuzumab (loading dose 8 mg/kg followed by a maintenance dose of 6 mg/kg) on day 1 and pertuzumab (loading dose 840 mg followed by a maintenance dose of 420 mg) on day 1, every 21 days as one cycle.

Surgery will be performed after completion of neoadjuvant chemotherapy, with intraoperative excision of specimens (breast + axilla) for pathological evaluation.

Comparative analysis of pCR, EFS, iDFS and safety outcomes between the two groups will be conducted using appropriate statistical methods.

Safety evaluation will include the incidence of adverse events, incidence of serious adverse events, dose adjustment rate, and discontinuation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years;
2. Clinical T2-T4d, or T1c with axillary lymph node positivity;
3. Histopathologically confirmed HER2-positive invasive breast cancer; Note: HER2 positivity was determined by immunohistochemical (IHC) staining of 3+ or, if IHC 2+, by HER2 gene amplification as demonstrated by fluorescence in situ hybridization (FISH) assay；
4. Have clinically measurable lesions: Measurable lesions shown on ultrasound, mammography, or MR (optional) within 1 month before randomization;
5. No chemotherapy contraindications detected by organ and bone marrow function tests within 1 month before chemotherapy:

   1. Neutrophil count absolute value ≧2.0×109/L;
   2. Hemoglobin ≧ 100g/L;
   3. Platelet count ≧100×109/L;
   4. Total bilirubin <1.5 ULN (upper limit of normal);
   5. Creatinine < 1.5×ULN
   6. AST/ALT < 1.5×ULN;
6. Cardiac ultrasound: Left ventricular ejection fraction (LVEF ≥ 55%);
7. Reproductive age women, negative serum pregnancy test within 14 days before randomization;
8. ECOG score 0 or 1;
9. Signature of informed consent.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Bilateral breast cancer;
3. Patients who have received chemotherapy, endocrine therapy, targeted therapy, or radiotherapy for this disease;
4. Patients with a second primary malignancy, except for adequately treated skin cancer;
5. Major non-breast cancer-related surgical procedures within the past 4 weeks before enrollment, or patients have not fully recovered from such surgical procedures;
6. Severe heart disease or conditions that do not allow participation in the study, including but not limited to the following:

   1. History of heart failure or systolic dysfunction (LVEF < 50%);
   2. High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher-grade atrioventricular conduction blocks (i.e., Mobitz II second-degree atrioventricular block or third-degree atrioventricular block);
   3. Angina pectoris requiring anti-anginal drug therapy;
   4. Clinically significant valvular heart disease;
   5. ECG showing a transmural myocardial infarction;
   6. Uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg);
7. Due to severe and uncontrolled other medical conditions, the investigator considers chemotherapy to be contraindicated;
8. Known history of allergy to any component of the study drugs; patients with a history of immune deficiency diseases, including HIV positivity, or patients with other acquired or congenital immune deficiency diseases, or a history of organ transplantation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | through study completion, an average of 1 year
  Pathological Complete Response (pCR) rate: It refers to the absence of any invasive cancer in the resected specimens (breast + axilla) after completion of neoadjuvant chemotherapy and surgery (i.e., ypT0/is, ypN0).

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5 years after surgery
  EFS is defined as the time from randomization to any of the following events: disease progression during neoadjuvant treatment, disease recurrence, or any cause of death.
Invasive Disease-Free Survival (iDFS) | 5 years after surgery
  This refers to the time from surgery to the first documented occurrence of an event such as ipsilateral invasive breast tumour recurrence, distant recurrence, contralateral invasive breast cancer, or death from any cause.
Safety-Number of adverse events and serious adverse events. | After each cycle of chemotherapy (21 days as 1 cycle)
  Safety will be assessed by evaluating the nature, incidence, and severity of chemotherapy-related adverse events according to CTCAE 4.0 (Common Terminology Criteria for Adverse Events).
Tolerability-Dose adjustment rate and withdrawal rate of chemotherapy drugs | After the end of the 6th cycle of chemotherapy (21 days as 1 cycle)
  Tolerability will be assessed by evaluating the dose adjustment rate and discontinuation rate of chemotherapy drugs in both treatment regimens.
Exploratory endpoint - Differences in pCR rates between predefined subgroups and factors influencing pCR in the study population. | through study completion, an average of 1 year
  The differences in pCR rate between various predefined subgroups and the factors affecting pCR in the enrolled population will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Study Principal Investigator Henan Cancer Hospital
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Chen XC, Jiao DC, Qiao JH, Wang CZ, Sun XF, Lu ZD, Li LF, Zhang CJ, Yan M, Wei Y, Chen B, Feng YQ, Deng M, Ma MD, Plichta JK, He YW, Liu ZZ. De-escalated neoadjuvant weekly nab-paclitaxel with trastuzumab and pertuzumab versus docetaxel, carboplatin, trastuzumab, and pertuzumab in patients with HER2-positive early breast cancer (HELEN-006): a multicentre, randomised, phase 3 trial. Lancet Oncol. 2025 Jan;26(1):27-36. doi: 10.1016/S1470-2045(24)00581-3. Epub 2024 Nov 26. PMID 39612919